CLINICAL TRIAL: NCT06849401
Title: A Single-arm, Open Label Clinical Study to Evaluate the Safety and Efficacy of VGO-Cs01p in Patients With CD7-positive Relapsed/Refractory Acute T-lymphoblastic Leukemia
Brief Title: The Safety and Efficacy of VGO-Cs01p in Patients With CD7-positive Relapsed/Refractory Acute T-lymphoblastic Leukemia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hui Zhang, Chief Physician, Shanghai Children's Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VGO-Cs01p-001
Record Dates: First submitted 2025-02-21; First posted 2025-02-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-02

CONDITIONS: T-ALL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGO-Cs01p (Experimental): Up to three sequential VGO-Cs01p dose levels （4e7、1.2e8、3.6e8 CAR-NK cells/kg）are planned. Each subject will accept six doses of VGO-Cs01p
  Interventions: Biological: VGO-Cs01p

INTERVENTIONS:
Biological: VGO-Cs01p — Off-the-shelf NK cell products derived from human embryonic stem cells (hESCs)

SUMMARY:
To learn if the VGO-Cs01p can help to control CD7-positive relapsed/refractory acute T-lymphoblastic leukemia (R/R T-ALL) in children.

DETAILED DESCRIPTION:
This is a single-arm, open label, IIT clinical trial to evaluate the safety and efficacy of CD7 CAR NK cells in subjects with CD7-positive relapsed/refractory acute T-lymphoblastic leukemia (R/R T-ALL). 5~9 subjects plan to be enrolled. In this study, safety and efficacy results will be used for dose escalation design at the same time, and three initial dose groups are set up. All subjects will be followed up to 12 months after infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥2 and ≤18 years old, male or female;
2. Subjects who have relapse or refractory T-cell lymphoblastic leukemia (T-ALL) according to the standards of the NCCN Clinical Practice Guidelines for Acute Lymphoblastic Leukemia (2024.V6);
3. Meets the criteria for recurrent or refractory T-ALL, including: a) Recurrent: Reappearance of blasts in peripheral blood or bone marrow (>25%) after complete remission or occurrence of extramedullary disease, and ineffectiveness of other treatments； b) Primary Refractory: Appearance of blasts in bone marrow ≥5% after 2 months standard induction chemotherapy, and no other treatment can be used as judged by the investigator;
4. After one cycle of other treatments (such as Olverembatinib combined with APG-125), the blasts remain≥5%;
5. Cell immunophenotyping confirmation of CD7 positive blasts >80%;
6. Estimated survival period >12 weeks;
7. Eastern Cooperative Oncology Group (ECOG) performance status score ≤1 or KPS > 60;
8. Left ventricular ejection fraction ≥50%;
9. Pulmonary function ≤ Grade 1 dyspnea (CTCAE v5.0), normal oxygen saturation without oxygen supplementation;
10. TBil ≤ 3×ULN, AST and ALT ≤ 5×ULN, creatinine ≤ 1.6 mg/dl within 1 week prior to enrollment;
11. Negative serum pregnancy test for fertile women; fertile non-abstinent female patients must agree to use an effective contraceptive method from screening to 1 year after cell infusion. Fertile male patients' partners must agree to use effective contraception from screening to 1 year after cell infusion, and should not donate semen or sperm throughout the study;
12. The subject or their legal guardian voluntarily participates in the study, understands the information, purpose, and risks described in the informed consent form, and can provide a signed and dated informed consent form;
13. The subject and/or their parents or their legal guardian should voluntary and able to comply with all requirements of the trial.

Exclusion Criteria:

1. Extramedullary involvement of the central nervous system or testicular at screening.
2. Patients with a history of severe CNS diseases, such as uncontrolled seizures, stroke, severe brain damage resulting in speech impairment, psychiatric disorders, etc;
3. NYHA functional class III or IV heart failure;
4. Presence of disseminated intravascular coagulation;
5. Presence of severe autoimmune diseases or immune deficiency diseases;
6. Active GVHD requiring systemic treatment;
7. Presence of other severe diseases, presence of gastrointestinal ulcers or active gastrointestinal bleeding, currently undergoing anticoagulant or antiplatelet therapy, or judged by the investigator to pose unacceptable surgical or anesthesia risks;
8. Currently receiving systemic steroids or other immunosuppressive therapy prior to screening, and still need long-term use after enrollment as judged by the investigator (excluding inhaled or local use);
9. History or concurrent active malignant tumors within 3 years prior to enrollment;
10. Active HBV or HCV infection (HBV-DNA positive or HCV-RNA positive), HIV positive, or positive syphilis test;
11. Other severe or persistent active infections;
12. Adverse events related to previous systemic immunotherapy (including other investigational drugs or medical device interventions) prior to enrollment have not reduced to grade 1 severity or returned to baseline;
13. Platelet count remains low after intervention treatment (meeting clinical transfusion criteria) prior to enrollment；
14. Discontinuation of immunosuppressive agents for less than 2 weeks;
15. Participation in CAR-T cell therapy or gene therapy at any time prior to screening;
16. History of allergy to any component of the study product;
17. Vaccination or any surgery within the 4 weeks prior to screening;
18. Other situations as judged by the investigator may increase the subject's risk or interfere with study;
19. Pregnant or breastfeeding women;
20. Individuals assessed by the investigator to have potential hidden risks of disputes.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 1 year post the first VGO-Cs01p infusion
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.

SECONDARY OUTCOMES:
ORR（Objective response rate） | 28 days and 1 year post the first VGO-Cs01p infusion
  Includes CR (complete response)/ CRh (CR with partial hematological recovery) /CRi (CR with incomplete hematological recovery)/PR（partial response）.
MRD (Minimal/Measurable Residual Diseas) | 1 year post the first VGO-Cs01p infusion
  Minimal/Measurable Residual Disease negative response rate
DOR (Duration of response) | 1 year post the first VGO-Cs01p infusion
  DOR is defined as the time from the first assessment of CR/CRh/CRi to relapse or death in clinical remission.
LFS (Leukemia-Free Survival) | 1 year post the first VGO-Cs01p infusion
  Defined as the time from clinical remission (CR/CRh/CRi) to relapse or death in clinical remission.
OS (Overall survival) | 1 year post the first VGO-Cs01p infusion
  Overall survival was defined as the time from the first infusion until the subject died or lost to follow-up for any cause.
PK parameters of VGO-Cs01p | 1 year post the first VGO-Cs01p infusion
  Cmax
Absolute value of CD7+ cells in peripheral blood | 1 year post the first VGO-Cs01p infusion
  PD parameters
Immunogenicity | 1 year post the first VGO-Cs01p infusion
  The number of subjects with antibodies to VGO-Cs01p and the antibody titer.
PK parameters of VGO-Cs01p | 1 year post the first VGO-Cs01p infusion
  Tmax
PK parameters of VGO-Cs01p | 1 year post the first VGO-Cs01p infusion
  AUC0-28
Proportion of CD7+ cells in peripheral blood | 1 year post the first VGO-Cs01p infusion
  PD parameters

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGO-Cs01p is fully approved.